CLINICAL TRIAL: NCT00975156
Title: Improving Ambulation Post Stroke With Robotic Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Elizabeth Noser, Clinical Assistant Professor - Neurology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MH-08-0206; Medallion Grant
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2012-09-13 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lokomat Intervention (Experimental): Lokomat gait training (five days a week for eight weeks for a total of 40 sessions).
  Interventions: Device: Lokomat
- Standard of Care (Active Comparator): Conventional physical therapy focusing on gait training for five days a week for eight weeks for a total of 40 sessions.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Conventional physical therapy
  Arms: Standard of Care
Device: Lokomat — Robotic-assisted walking device
  Arms: Lokomat Intervention

SUMMARY:
The purpose of this research study is to look at a new rehabilitation technique for individuals who have suffered a stroke and have difficulties walking. This study is designed to compare robot-assisted (Lokomat) rehabilitation therapy with standard physical therapy in order to improve walking post-stroke. This research project will be conducted as a pilot randomized controlled trial that compares the effectiveness of Lokomat versus conventional physical therapy in improving the ambulation and gait of chronic stroke patients. The project will provide important pilot data that could indicate whether or not the effectiveness of Lokomat training is superior to that of standard physical therapy and if a definitive and larger clinical trial is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ischemic or hemorrhagic stroke confirmed by cerebral computed tomography (CT) or magnetic resonance imaging (MRI) scan
* Age>18
* At least 3 months post stroke at time of enrollment into study
* Ability to walk at least 10 feet with maximum 1 person assist, but not to walk in the community independently
* Residual paresis in the lower extremity as defined by the National Institute of Health Stroke Scale lower extremity motor score 2-4
* Ability to perform Lokomat ambulation training with assistance of 1 therapist
* Ability to follow a three-step command
* Physician approval for patient participation
* Ability to give informed consent
* Completed their rehabilitation services, i.e., receiving no concurrent physical, occupational, or speech therapies

Exclusion Criteria:

* Serious cardiac condition
* Uncontrolled blood pressure, defined as > 200 or diastolic > 100 at rest
* Hx of serious chronic obstructive pulmonary disease or oxygen dependence
* Sever weight bearing pain
* Lower extremity amputation
* Claudication while walking
* Life expectancy < 1 year
* History of deep vein thrombosis/pulmonary embolism (DVT/PE) within 6 months
* Severe orthopedic problem
* Any medical or psychiatric condition that the investigators believe would make the patient unable to participate in this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Noser, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Conventional physical therapy
Period: Overall Study
Arm/Group | Lokomat Intervention | Standard of Care
Started | 11 | 10
Completed | 11 | 9
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lokomat Intervention | Standard of Care | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 7 | 5 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 66.91 (8.50) | 64.33 (10.91) | 65.75 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: 10-meter Walking Test (10mWT)
Time Frame: Baseline, 1 Week Post-Intervention (study mean of 5.05 days since last therapy session), 3-Month Post-Intervention
Population: Analysis was determined per protocol (i.e.between-group variation)
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Groups:
- Lokomat Intervention 10-meter Walking Test (10mWT) Outcome; Standard of Care 10mWT Outcome; All Participants 10mWT Outcome: Baseline, 1-Week Post-Intervention (study mean of 5.05 days since last therapy session), 3-Month Post-Intervention assessment values measured by a blinded assessor.
Arm/Group | Lokomat Intervention 10-meter Walking Test (10mWT) Outcome | Standard of Care 10mWT Outcome | All Participants 10mWT Outcome
Number analyzed (Participants) | 11 | 9 | 20
meters per second (m/s)
  Baseline | 0.20 (0.10) | 0.18 (0.12) | 0.19 (0.11)
  Post-Intervention (mean=5.05 days post-therapy) | 0.20 (0.10) | 0.27 (0.27) | 0.23 (0.19)
  Three-Month Follow-up | 0.21 (0.10) | 0.28 (0.29) | 0.24 (0.20)

2. Secondary Outcome: 6 Minute Walking Distance (6MWD)
Time Frame: Baseline, 1-Week Post-Intervention (study mean of 5.05 days since last therapy session), 3-Month Post-Intervention
Measure: Mean (Standard Deviation); unit: meters (m)
Groups:
- Lokomat Intervention 6 Minute Walking Distance (6MWD) Outcome; Standard of Care 6MWD Outcome: Baseline, 1-Week Post-Intervention (study mean of 5.05 days since last therapy session), 3-Month Post-Intervention assessments were completed by a blinded assessor.
- All Participants 6MWD Outcome: Baseline, Post-Intervention (study mean of 5.05 days since last therapy session), 3-Month Post-Intervention assessments were completed by a blinded assessor.
Arm/Group | Lokomat Intervention 6 Minute Walking Distance (6MWD) Outcome | Standard of Care 6MWD Outcome | All Participants 6MWD Outcome
Number analyzed (Participants) | 11 | 9 | 20
meters (m)
  Baseline | 53.94 (30.53) | 48.77 (21.04) | 51.61 (26.16)
  Post-Intervention (mean=5.05 days post-therapy) | 57.02 (25.50) | 70.26 (60.40) | 62.98 (43.86)
  Three-Month Follow-up | 57.82 (25.99) | 76.89 (62.29) | 66.40 (45.65)

ADVERSE EVENTS:
Groups:
- Lokomat Intervention: Robotic-assisted gait therapy
Arm/Group | Lokomat Intervention | Standard of Care
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/9
Other Adverse Events (participants affected / at risk) | 5/11 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lokomat Intervention (N=11) | Standard of Care (N=9)
Skin breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin breakdown as a result of therapy; adverse event deemed "definitely related" to protocol.
Hypotensive episode (Cardiac disorders) | 0 (0) | 1 (1) — Sudden drop in blood pressure at subject's home leading to brief hospitalization; adverse event deemed "unrelated" to protocol.
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) — Sudden chest pain prior to therapy leading to ER visit and brief hospitalization; adverse event deemed "unrelated" to protocol.
Stroke (Vascular disorders) | 1 (1) | 0 (0) — Subject with a second stroke during the post-treatment phase of study participation; adverse event deemed "unrelated" to protocol.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lokomat Intervention (N=11) | Standard of Care (N=9)
Minor skin breakdown (Skin and subcutaneous tissue disorders) | 5 (12) | 3 (3) — minor skin breakdown

LIMITATIONS AND CAVEATS:
Limitations include: small sample (n=21 enrolled, n=20 completed) and significant (p=0.025) difference between groups in time since stroke (Lokomat group, time since stroke mean=1353.60 days; Conventional group, time since stroke mean=525.00 days).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No